CLINICAL TRIAL: NCT06006104
Title: A Phase I/II Clinical Study to Evaluate the Pharmacokinetics, Radiation Dosimetry, Safety and Preliminary Efficacy of HRS-4357 in Patients With PSMA Positive Advanced Prostate Cancer
Brief Title: Phase 1/2 Clinical Study of HRS-4357 in Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4357-101
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-4357 injection (Experimental)
  Interventions: Drug: HRS-4357 injection

INTERVENTIONS:
Drug: HRS-4357 injection — HRS-4357 injection

SUMMARY:
The study is being conducted to evaluate the the safety, pharmacokinetics, radiation dosimetry, and preliminary efficacy of HRS-4357 injection in adult patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this clinical trial, understanding of the study procedures and being able to sign the informed consent form in writing;
2. Male, age ≥18 years;
3. ECOG score 0 - 1;
4. Histologically and/or cytologically confirmed adenocarcinoma of the prostate;

Exclusion Criteria:

1. Spinal cord compression with clinical symptoms, or clinical symptoms and/or imaging findings suggesting imminent spinal cord compression.
2. Severe urinary incontinence, hydronephrosis, severe micturition dysfunction, etc. Note: Subjects with bladder outflow obstruction or urinary incontinence that can be controlled by the best available standard of care (including pads, drainage, etc.) are eligible to participate in the study.
3. Active syphilis infection.
4. Known hypersensitivity to components of the study drug or its analogues.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Prog Dose limiting toxicity (DLT) | up to 9 months follow-up
recommended phase 2 dose (RP2D) | up to 9 months follow-up
recommended dosing cycle. | up to 9 months follow-up
PSA50 response rate | up to 12 weeks follow-up

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 6 weeks follow-up
time to maximum plasma concentration (Tmax) | up to 6 weeks follow-up
area under the plasma concentration-time curve (AUC) | up to 6 weeks follow-up
clearance (Cl) | up to 6 weeks follow-up
volume of distribution (Vz) | up to 6 weeks follow-up
terminal half-life (t1/2) | up to 6 weeks follow-up
cumulative urinary excretion of radioactive dose | up to 6 weeks follow-up
Absorbed dose and effective dose of radioactive internal irradiation of the whole body and major organs; | up to 6 weeks follow-up
PSA90 response rate | up to 12 weeks follow-up]
time to PSA progression | up to 9 months follow-up
Overall Response Rate (ORR) | up to 20 months follow-up
Disease control Rate (DCR) | up to 20 months follow-up
Duration of Response (DoR) | up to 20 months follow-up
Radiographic Progression-free Survival (rPFS) | up to 9 months follow-up
Overall Survival (OS) | up to 20 months follow-up
Incidence and severity of AEs and SAEs | up to 20 months follow-up

IPD SHARING:
Plan to Share IPD: Undecided